CLINICAL TRIAL: NCT06818136
Title: Evaluation of the Efficacy of Bladder EpiCheck® for the Primary Detection of Urothelial Carcinoma in Subjects Presenting With Haematuria
Brief Title: Bladder EpiCheck European Haematuria Study
Status: Recruiting | Type: Observational
Sponsor: Nucleix Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 68096
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hematuria; Cystoscopy; Urothelial Carcinoma Bladder; Urothelial Carcinoma of the Renal Pelvis and Ureter; Urothelial Carcinoma of the Urinary Bladder
Keywords: urine test; methylation; primary detection
MeSH Terms: conditions — Hematuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — voided urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- aged ≥ 45 years with haematuria scheduled for cystoscopy, for suspicion of urothelial carcinoma: Adult participants aged ≥ 45 years presenting with haematuria in the past 6 months, scheduled to undergo haematuria workup, including cystoscopy, for suspicion of urothelial carcinoma.
  Interventions: Diagnostic Test: Bladder EpiCheck

INTERVENTIONS:
Diagnostic Test: Bladder EpiCheck — The participant will provide a voided urine sample, which will be tested using the Bladder EpiCheck test. The clinical care team and the participant will not be informed of the result, and the standard of care will not change.

SUMMARY:
The goal of this observational study is to further validate the sensitivity and specificity of Bladder EpiCheck in primary detection of urothelial carcinoma in participants aged 45 years or older presenting with haematuria, compared to cystoscopy and pathology, if performed.

Participants will provide a voided urine sample, and data from standard of care haematuria work-up will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 45 years or older
2. Participants who are willing and able to provide written informed consent and adhere to study procedures
3. Participants presenting with visible and/or non-visible haematuria within 6 months prior to study enrollment
4. Participants scheduled to undergo standard of care cystoscopy for urinary bladder examination within 60 days after study enrollment
5. Participants who are able to produce at least 10 ml of voided urine

Exclusion Criteria:

1. Participants with history of urothelial cancer in the bladder and/or upper urinary tract
2. Participants who had prior cystoscopy for haematuria within the past 2 years
3. Participants previously enrolled in this study
4. Participants treated for prostate cancer within the last 12 months
5. Participants treated for kidney cancer within the last 12 months
6. Participants with untreated urinary tract infection
7. Participants with symptomatic urinary tract stones (e.g. flank pain)
8. Participants on dialysis for end stage renal failure
9. Participants with a long term urinary catheter
10. Pregnancy (self-reported)
11. Participants who, because of medical status, or frailty is not expected to be able to complete the full diagnostic pathway

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: aged ≥ 45 years with haematuria scheduled for cystoscopy, for suspicion of urothelial carcinoma
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of Bladder EpiCheck to detect primary urothelial carcinoma | urothelial carcinoma detected within 6 months of enrolment, by the standard of care haematuria work-up
  The sensitivity and specificity of Bladder EpiCheck to detect primary urothelial carcinoma, calculated versus the Reference Standard defined by cystoscopy, imaging, and, if indicated, pathological confirmation) in participants presenting with haematuria (visible and/or non-visible).

SECONDARY OUTCOMES:
Non-inferiority of Bladder EpiCheck overall sensitivity vs. cytology in detection of primary urothelial carcinoma | urothelial carcinoma detected within 6 months of enrolment, by the standard of care haematuria work-up
Non-inferiority of Bladder EpiCheck specificity vs. cytology in detection of primary urothelial carcinoma | urothelial carcinoma detected within 6 months of enrolment, by the standard of care haematuria work-up
Further validate the sensitivity of the Bladder EpiCheck test to detect pathologically confirmed high-grade urothelial carcinoma, including HG non-muscle invasive and muscle invasive disease. | urothelial carcinoma detected within 6 months of enrolment, by the standard of care haematuria work-up

CONTACTS AND LOCATIONS:
Overall Officials: Paramananthan Mariappan, MB BS PhD FRCS(Urol) FEBU FRCS, Principal Investigator — Western General Hospital, Edinburgh
Locations (5):
- United Kingdom (5):
  - NHS Fife, Dunfermline, Fife
  - Addenbrooke's Hospital, Cambridge
  - NHS Lothian, Edinburgh
  - Guy's and St Thomas, London
  - Frimley, Surrey Quays

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Witjes JA, Morote J, Cornel EB, Gakis G, van Valenberg FJP, Lozano F, Sternberg IA, Willemsen E, Hegemann ML, Paitan Y, Leibovitch I. Performance of the Bladder EpiCheck Methylation Test for Patients Under Surveillance for Non-muscle-invasive Bladder Cancer: Results of a Multicenter, Prospective, Blinded Clinical Trial. Eur Urol Oncol. 2018 Sep;1(4):307-313. doi: 10.1016/j.euo.2018.06.011. Epub 2018 Jul 17. PMID 31100252